CLINICAL TRIAL: NCT04990271
Title: A Clinical Study on the Efficacy and Safety of VEC Intravenous Chemotherapy Combined With Conbercept Intravitreal Injection in the Treatment of Retinoblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V2.3
Record Dates: First submitted 2021-07-23; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma; Conbercept; VEC Intravenous Chemotherapy
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Conbercept intravitreal Injection (Experimental)
  Interventions: Drug: Conbercept ophthalmic injection

INTERVENTIONS:
Drug: Conbercept ophthalmic injection — Monthly injection of Conbercept from 0~5 months
  Other Names: KH902

SUMMARY:
This prospective, multi-center, open single-arm Phase II clinical trial is designed to investigate the efficacy and safety of intravenous chemotherapy combined with Conbercept intravitreal injection in the treatment of retinoblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's guardian signs an informed consent form and is willing to receive follow-up according to the schedule of the trial;
2. Children of more than 3 months and under 5 years of age who have not received any anti-cancer treatment;
3. The target eye must meet the following requirements:

   Clinically diagnosed as monocular retinoblastoma; According to the IIRC diagnostic criteria, the treatment eye is classified as Group E stage without clinical high-risk factors (Table 1); No refractive medium turbidity and/or pupillary abnormalities that affect the fundus examination; IOP≤21mmHg.
4. Sufficient organ function at baseline.

Exclusion Criteria:

Subjects with any of the following eye conditions:

1. Patients diagnosed as stage E retinoblastoma in one eye, but with high-risk factors: neovascular glaucoma; refractive interstitial opacity caused by anterior chamber, vitreous or subretinal hemorrhage; tumor invasion of optic nerve posterior to the cribriform plate and choroid (range of diameter> 2 mm), sclera, and anterior chamber;
2. Treatment-naïve pediatric patients;

Patients with any of the following systemic diseases:

1. With a history of allergies or have allergic reactions to fluorescein sodium, with a history of allergies to protein products for treatment or diagnosis, and have allergic reactions to two or more drugs and/or non-drug factors, or suffering from allergic diseases;
2. Low birth weight children, and severely growth-stunted children;
3. Children who need systemic treatment for other system diseases;
4. Any condition that should be excluded from the study in the opinion of the investigator.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the 1-year ocular salvage rate of intravenous chemotherapy combined with Conbercept intravitreal injection in the treatment of retinoblastoma | 1 year
  12-month ocular salvage rate: calculate the number and percentage of subjects who reach 12-month ocular salvage rate, and use the exact probability method to estimate 95% CI.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Henan Children's Hospital, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No